CLINICAL TRIAL: NCT02867943
Title: Effects of Respiratory Rate on Venous-to-arterial CO2 Tension Difference in Septic Shock Patients Under Volume Mechanical Ventilation
Brief Title: GapCO2 and Respiratory Rate in Patients Under Volume Mechanical Ventilation
Acronym: gapCO2
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: 105 Hospital of Chinese People's Liberation Army (Other)
Responsible Party: Sponsor
Other Study IDs: PLA-105-ICU
Record Dates: First submitted 2016-08-11; First posted 2016-08-16 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-08

CONDITIONS: Shock
Keywords: sepsis, shock,Lactate,volume controlled ventilation
MeSH Terms: conditions — Shock; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- respiratory rate is 10 breaths/min: GapCO2=Pv-aCO2 = PvCO2 - PaCO2;
  Effects of venous-to-arterial CO2 tension difference after increased respiratory rate.
  Interventions: Other: Effects of respiratory rate on gapCO2
- respiratory rate is 12 breaths/min: GapCO2=Pv-aCO2 = PvCO2 - PaCO2;
  Effects of venous-to-arterial CO2 tension difference after increased respiratory rate.
  Interventions: Other: Effects of respiratory rate on gapCO2
- respiratory rate is 14 breaths/min: GapCO2=Pv-aCO2 = PvCO2 - PaCO2;
  Effects of venous-to-arterial CO2 tension difference after increased respiratory rate.
  Interventions: Other: Effects of respiratory rate on gapCO2
- respiratory rate is 16 breaths/min: GapCO2=Pv-aCO2 = PvCO2 - PaCO2;
  Effects of venous-to-arterial CO2 tension difference after increased respiratory rate.
  Interventions: Other: Effects of respiratory rate on gapCO2

INTERVENTIONS:
Other: Effects of respiratory rate on gapCO2 — respiratory rate was started at 10 breaths/min and added by 2 breaths/min every 60 min up to 16 breaths/min

SUMMARY:
As an approximate of the difference between venous-to-arterial CO2 tension (∆PCO2), ∆PCO2 is proportional to CO2 production and inversely related to cardiac output (Fick equation). Anaerobic CO2 production is thought to occur when tissue hypoxia is present, mostly because of buffering of bicarbonate ions by the protons produced in excess secondary to the hydrolysis of adenosine triphosphate. Therefore ∆PCO2 has been proposed as a marker of tissue hypoxia.

DETAILED DESCRIPTION:
An increased ∆PCO2 (> 6 mmHg) could be used to identify patients who still remain inadequately resuscitated, when deciding when to continue resuscitation despite a central venous oxygen saturation (ScvO2) > 70% associated with elevated blood lactate levels.

Under steady states of both VO2 and VCO2, P (v-a) CO2 was observed to increase in parallel with the reduction in cardiac output. However, spontaneous breathing and hyperventilation may reduce PaCO2 and prevent the CO2 stagnation-induced rise in PvCO2.

To date,these studies of ∆PCO2 and respiratory rate in septic shock patients Under Volume Mechanical Ventilation are rarely.

ELIGIBILITY:
Inclusion Criteria:

Patients were included in the study, if the attending physician find the persistence of signs of hypoperfusion (oliguria, mottled skin, central venous oxygen saturation (ScvO2) <70 % despite a hemoglobin > 8 g/dl),despite achieving adequate intravascular volume and adequate mean arterial pressure (MAP) > 65 mmHg as recommended by the Surviving Sepsis Campaign.

Exclusion Criteria:

Exclusion criteria were pregnancy, COPD，age less than 18 years old, unstable hemodynamic condition (change of vasoactive drug dosage or fluid administration within 1 h preceding the protocol) and uncontrolled tachyarrhythmias (heart rate>140 beats/min).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects were sequentially admitted to the Department of Critical Care Medicine of 105 Hospital of PLA from March of 2016 till the end of this study.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-10 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Effects of respiratory rate on venous-to-arterial CO2 tension difference in septic shock patients Under Volume Mechanical Ventilation | 1 year

IPD SHARING:
Plan to Share IPD: Yes